CLINICAL TRIAL: NCT01691326
Title: Safety and Immunogenicity Among Healthy Children Receiving Fluzone® Influenza Virus Vaccine (2012-2013 Formulation)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRC49; U1111-1124-8218 (Other: WHO)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® (Influenza Virus Vaccine) 2012-2013 Formulation; Influenza virus vaccine; Trivalent Inactivated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 months to < 36 months of age group (Experimental): Participants at 6 months to < 36 months of age at the time of enrollment will receive Influenza Virus Vaccine, No Preservative; Fluzone® (Pediatric Dose).
  Interventions: Biological: Fluzone®: Influenza Virus Vaccine, No Preservative: Pediatric Dose
- 3 years to < 9 years of age group (Experimental): Participants at 3 years to < 9 years of age at the time of enrollment will receive Influenza Virus Vaccine, No Preservative; Fluzone®.
  Interventions: Biological: Fluzone®; Influenza Virus Vaccine, No Preservative

INTERVENTIONS:
Biological: Fluzone®: Influenza Virus Vaccine, No Preservative: Pediatric Dose — 0.25 mL dose, Intramuscular
  Other Names: Fluzone® (Influenza Virus Vaccine) 2012-2013 Formulation
  Arms: 6 months to < 36 months of age group
Biological: Fluzone®; Influenza Virus Vaccine, No Preservative — 0.5 mL dose, Intramuscular
  Other Names: Fluzone® (Influenza Virus Vaccine) 2012 2013 Formulation
  Arms: 3 years to < 9 years of age group

SUMMARY:
The aim of this clinical study is to demonstrate safety and immunogenicity of Fluzone vaccine.

Objective:

* To describe the safety of the 2012-2013 formulation of Fluzone vaccine, administered in a 1- or 2-dose schedule, in accordance with Advisory Committee on Immunization Practices (ACIP) recommendations, in children 6 months to < 9 years of age.

Observational Objectives:

* To describe the immunogenicity of the 2012-2013 formulation of Fluzone vaccine, administered in a 1- or 2-dose schedule in accordance with ACIP recommendations, in children 6 months to < 9 years of age.
* To submit remaining available sera from subjects to the Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), the Centers for Disease Control and Prevention (CDC), and the Food and Drug Administration (FDA) to support selection and recommendation of strains for subsequent years' influenza vaccines.

DETAILED DESCRIPTION:
All participants will receive Fluzone vaccine during Visit 1. For subjects receiving 2 doses of influenza vaccine, per ACIP guidance, a second dose of Fluzone vaccine will be administered during Visit 2.

Total duration of participation in the study is approximately 28 days for participants receiving 1 dose and 56 days for those receiving 2 doses of Fluzone vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 6 months to < 9 years of age on the day of inclusion
* Parent/guardian is willing and able to attend scheduled visits and to comply with the study procedures during the entire duration of the study
* Assent form has been signed and dated by subjects 7 to < 9 years of age, and informed consent form has been signed and dated by parent(s) or another legally acceptable representative
* For subjects 6 months to < 24 months of age, born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg (5.5 lbs).

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, latex, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Prescribing Information)
* History of serious adverse reaction to any influenza vaccine
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before Visit 2 for subjects receiving 1 influenza vaccine or Visit 3 for subjects receiving 2 doses of influenza vaccine
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study
* Prior vaccination with any formulation of 2012-2013 influenza vaccine
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator
* Thrombocytopenia, which may be a contraindication for IM vaccination, at the discretion of the Investigator
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine
* Personal history of Guillain-Barré syndrome
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Known seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4°F). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Identified as a natural or adopted child of the Investigator or an employee with direct involvement in the proposed study.

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- United States (2):
  - Bardstown, Kentucky
  - Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 19 September 2012 to 12 December 2012 at 2 clinic centers in the United States.
Pre-assignment Details: A total of 60 participants who met all of the inclusion and none of the exclusion criteria were randomized and vaccinated in this study.
Groups:
- Age 6 to < 36 Months Group: Participants 6 months to < 36 months of age that received one or two doses of 0.25 mL of Fluzone vaccine
- Age 3 to < 9 Years Group: Participants 3 years to < 9 years of age that received one or two doses 0.5 mL of Fluzone vaccine
Period: Overall Study
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age 3 to < 9 Years Group: Participants 3 years to < 9 years of age that received one or two doses of 0.5 mL of Fluzone vaccine
- Total: Total of all reporting groups
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 60
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.8 (0.6) | 5.2 (1.6) | 3.5 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions Following Vaccination With Fluzone® Influenza Virus Vaccine (2012-2013 Formulation)
Description: Solicited injection site reactions (Age 6 to < 24 Months): Tenderness, Erythema and Swelling. Solicited systemic reactions: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite, and Irritability.
  Grade 3: Tenderness, Cries when injected limb is moved; Erythema and Swelling, ≥ 50 mm; Fever, >103.1°F; Vomiting, ≥6 episodes/24 hours; Abnormal crying, >3 hours; Drowsiness, Sleeping most of the time; Loss of appetite, Refuses ≥3 feeds/meals or most feeds/meals; Irritability, Inconsolable.
  Solicited injection site reactions (Age 24 Months to < 9 Years): Pain, Erythema, and Swelling. Systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia.
  Grade 3: Pain, Incapacitating, unable to perform usual activities; Redness and Swelling, ≥ 50 mm; Fever: ≥102.1°F; Headache, Malaise, and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed using the Safety Analysis Set, which includes all persons who received at least one dose of study vaccine.
Measure: Number; unit: Participants
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group
Number analyzed (Participants) | 30 | 30
Participants
  Injection site Tenderness (N = 15, 0) | 8 | NA [0 to 0] — Injection site Tenderness was not solicited in this group
  Grade 3 Injection site Tenderness (N =15, 0) | 1 | NA [0 to 0] — Injection site Tenderness was not solicited in this group
  Injection site Pain (N =15, 30) | 8 | 13 [0 to 0]
  Grade 3 Injection site Pain (N = 15, 30) | 0 | 0 [0 to 0]
  Injection site Erythema (N = 30, 30) | 8 | 9 [0 to 0]
  Grade 3 Injection site Erythema (N = 30, 30) | 0 | 0 [0 to 0]
  Injection site Swelling (N = 30, 30) | 5 | 7 [0 to 0]
  Grade 3 Injection site Swelling (N = 30, 30) | 0 | 0 [0 to 0]
  Fever (N = 30, 28) | 2 | 0 [0 to 0]
  Grade 3 Fever (N = 30, 28) | 0 | 0 [0 to 0]
  Headache (N = 15, 30) | 1 | 5 [0 to 0]
  Grade 3 Headache (N = 15, 30) | 0 | 0 [0 to 0]
  Malaise (N = 15, 30) | 4 | 4 [0 to 0]
  Grade 3 Malaise (N = 15, 30) | 0 | 0 [0 to 0]
  Myalgia (N = 15, 30) | 3 | 2 [0 to 0]
  Grade 3 Myalgia (N = 15, 30) | 0 | 0 [0 to 0]
  Vomiting (N = 15, 0) | 1 | NA [0 to 0] — Vomiting was not solicited in this group
  Grade 3 Vomiting (N = 15, 0) | 0 | NA [0 to 0] — Vomiting was not solicited in this group
  Abnormal crying (N = 15, 0) | 6 | NA [0 to 0] — Abnormal crying was not solicited in this group
  Grade 3 Abnormal crying (N = 15, 0) | 0 | NA [0 to 0] — Abnormal crying was not solicited in this group
  Drowsiness (N = 15, 0) | 5 | NA [0 to 0] — Drowsiness was not solicited in this group
  Grade 3 Drowsiness (N = 15, 0) | 0 | NA [0 to 0] — Drowsiness was not solicited in this group
  Loss of Appetite (N = 15, 0) | 4 | NA [0 to 0] — Loss of Appetite was not solicited in this group
  Grade 3 Loss of Appetite (N = 15, 0) | 0 | NA [0 to 0] — Loss of Appetite was not solicited in this group
  Irritability (N = 15, 0) | 9 | NA [0 to 0] — Irritability was not solicited in this group
  Grade 3 Irritability (N = 15, 0) | 1 | NA [0 to 0] — Irritability was not solicited in this group

2. Other Pre Specified Outcome: Geometric Mean Titers of Antibodies to Influenza Antigens Before and Following Vaccination With Fluzone® Influenza Virus Vaccine (2012-2013 Formulation).
Description: The influenza virus antibodies were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Geometric mean titers of antibodies against the influenza virus antigens were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- 6 to < 36 Months Age Group: Participants 6 months to < 36 months of age that received one or two doses of 0.25 mL of Fluzone vaccine
- 3 to < 9 Years Age Group: Participants 3 years to < 9 years of age that received one or two doses of 0.5 mL of Fluzone vaccine
Arm/Group | 6 to < 36 Months Age Group | 3 to < 9 Years Age Group
Number analyzed (Participants) | 25 | 30
Titers
  A/H1N1 (pre-vaccination) | 20.6 [9.93 to 42.6] | 68.8 [30.5 to 155]
  A/H1N1 (post-vaccination) | 334 [189 to 589] | 864 [559 to 1337]
  A/H3N2 (pre-vaccination) | 23.3 [11.4 to 47.5] | 84.8 [49.5 to 145]
  A/H3N2 (post-vaccination) | 506 [296 to 865] | 895 [585 to 1369]
  B (pre-vaccination) | 5.82 [4.76 to 7.13] | 9.66 [7.42 to 12.6]
  B (post-vaccination) | 16.7 [11.2 to 24.8] | 69.6 [46.4 to 105]

3. Other Pre Specified Outcome: Number of Participants With Seroprotection Before and Following Vaccination With Fluzone® Influenza Virus Vaccine (2012-2013 Formulation)
Description: Influenza virus antibodies were measured using a HAI assay. Seroprotection was defined as a titer ≥40 (1/dilution).
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Seroprotection against the influenza virus antigens were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group
Number analyzed (Participants) | 25 | 30
Participants
  A/H1N1 (pre-vaccination) | 10 | 18 [0 to 0]
  A/H1N1 (post-vaccination) | 24 | 30 [0 to 0]
  A/H3N2 (pre-vaccination) | 11 | 20 [0 to 0]
  A/H3N2 (post-vaccination) | 25 | 30 [0 to 0]
  B (pre-vaccination) | 1 | 2 [0 to 0]
  B (post-vaccination) | 6 | 21 [0 to 0]

4. Other Pre Specified Outcome: Number of Participants With Seroconversion Against Influenza Virus Antigens Following Vaccination With Fluzone® Influenza Virus Vaccine (2012-2013 Formulation)
Description: Influenza virus antibodies were measured using a HAI assay. Seroconversion was defined as a pre-vaccination titer <10 (1/dilution) and a post-vaccination titer ≥40 (1/dilution), or a pre-vaccination titer ≥10 (1/dilution) and ≥4-fold increase in titer 28 days after final vaccination.
Time Frame: Day 28 after final vaccination
Population: Seroconversion against the influenza virus antigens were assessed in the Per-protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group
Number analyzed (Participants) | 25 | 30
Participants
  A/H1N1 | 22 | 22 [0 to 0]
  A/H3N2 | 23 | 25 [0 to 0]
  B | 5 | 20 [0 to 0]

5. Other Pre Specified Outcome: Geometric Mean Titer Ratios (GMTRs) of Antibodies to Influenza Virus Antigens Following Vaccination With Fluzone® Influenza Virus Vaccine (2012-2013 Formulation).
Description: Influenza virus antibodies were measured using a HAI assay. Geometric mean titer ratio is the geometric mean of the individual post-vaccination / pre-vaccination titer of antibodies to the influenza virus antigens
Time Frame: Day 0 (pre-vaccination) and Day 28 after final vaccination
Population: Geometric mean titer ratios against the influenza virus antigens were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Age 6 to < 36 Months Group | Age 3 to < 9 Years Group
Number analyzed (Participants) | 25 | 30
Ratio
  A/H1N1 | 11.6 [7.24 to 18.7] | 10.7 [5.56 to 20.5]
  A/H3N2 | 16.2 [9.45 to 27.9] | 10.3 [5.88 to 18.1]
  B | 1.82 [1.29 to 2.55] | 5.34 [3.75 to 7.60]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 after final vaccination.
Arm/Group | 6 to < 36 Months Age Group | 3 to < 9 Years Age Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 9/30 | 13/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 6 to < 36 Months Age Group (N=30) | 3 to < 9 Years Age Group (N=30)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Injection site Tenderness (General disorders) | 8/15 (8) | 0/0 (0)
Injection site Pain (General disorders) | 8/15 (8) | 13 (13)
Injection site Erythema (General disorders) | 8 (8) | 9 (9)
Injection site Swelling (General disorders) | 5 (5) | 7 (7)
Fever (General disorders) | 2 (2) | 0/28 (0)
Abnormal crying (Psychiatric disorders) | 6/15 (6) | 0/0 (0)
Drowsiness (Nervous system disorders) | 5/15 (5) | 0/0 (0)
Loss of Appetite (Metabolism and nutrition disorders) | 4/15 (4) | 0/0 (0)
Irritability (Psychiatric disorders) | 9/15 (9) | 0/0 (0)
Headache (Nervous system disorders) | 1/15 (1) | 5 (5)
Malaise (General disorders) | 4/15 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3/15 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1/15 (1) | 0/0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications